CLINICAL TRIAL: NCT01259297
Title: A Randomized Controlled Trial of Aliskiren in the Prevention of Major Cardiovascular Events in Elderly People
Acronym: APOLLO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early in agreement with Health Authorities for feasibility reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100G2301; 2009-010170-38 (EudraCT Number)
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Events
Keywords: Aliskiren; Elderly; Major Cardiovascular Events; Effect of aliskiren-based regimen on major CV events (composite of CV death, non-fatal MI, non-fatal stroke and significant heart failure) in the elderly
MeSH Terms: interventions — aliskiren; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- Aliskiren + Amlodipine (Experimental): In run-in period (4-5 weeks) , patients on thiazide background therapy and approximately 50% of patients on neither CCB nor thiazide background therapy received Amlodipine 5 mg and Aliskiren 150/300 mg daily in a titrated manner as per protocol.
  In double blind period, patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  Patients randomized to this arm received Aliskiren 300 mg + Amlodipine 5 mg once daily during the double blind period.
  Interventions: Drug: Aliskiren; Drug: Amlodipine
- Aliskiren + Hydrochlorothiazide (HCTZ) (Experimental): In run-in period (4-5 weeks) , patients on CCB background therapy and approximately 50% of patients on neither thiazide nor CCB background therapy: received Hydrochlorothiazide 12.5/25 mg and Aliskiren 150/300 mg daily in a titrated manner as per protocol.
  In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  Patients randomized to this arm received Aliskiren 300 mg + HCTZ 25 mg once daily.
  Interventions: Drug: Aliskiren; Drug: Hydrochlorothiazide (HCTZ)
- Aliskiren + Placebo for Amlodipine (Experimental): In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  In double blind period, randomized patients to this arm received Aliskiren 300 mg + Placebo for Amlodipine 5 mg
  Interventions: Drug: Aliskiren; Drug: Placebo for Amlodipine
- Aliskiren + Placebo for HCTZ (Experimental): In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  In double blind period, randomized patients to this arm received Aliskiren 300 mg + Placebo for HCTZ 25 mg once daily
  Interventions: Drug: Aliskiren; Drug: Placebo for Hydrochlorothiazide (HCTZ)
- Amlodipine + Placebo for Aliskiren (Experimental): In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  In double blind period, randomized patients to this arm received Amlodipine 5 mg + placebo for Aliskiren 300 mg once daily
  Interventions: Drug: Amlodipine; Drug: Placebo for Aliskiren
- HCTZ + Placebo for Aliskiren (Experimental): In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  In double blind period, randomized patients to this arm received HCTZ 25 mg + placebo for Aliskiren 300 mg once daily
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Placebo for Aliskiren
- Placebo for Aliskiren + Placebo for Amlodipine (Placebo Comparator): In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  In double blind period, randomized patients to this arm received placebo for Aliskiren 300 mg + placebo for Amlodipine 5 mg once daily
  Interventions: Drug: Placebo for Aliskiren; Drug: Placebo for Amlodipine
- Placebo for Aliskiren + Placebo for HCTZ (Placebo Comparator): In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  In double blind period, randomized patients to this arm received placebo for Aliskiren 300 mg + placebo for HCTZ 25 mg once daily
  Interventions: Drug: Placebo for Aliskiren; Drug: Placebo for Hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150/300 mg once daily
  Arms: Aliskiren + Amlodipine; Aliskiren + Hydrochlorothiazide (HCTZ); Aliskiren + Placebo for Amlodipine; Aliskiren + Placebo for HCTZ
Drug: Amlodipine — Amlodipine 5 mg
  Arms: Aliskiren + Amlodipine; Amlodipine + Placebo for Aliskiren
Drug: Hydrochlorothiazide (HCTZ) — HCTZ 12.5/25 mg
  Arms: Aliskiren + Hydrochlorothiazide (HCTZ); HCTZ + Placebo for Aliskiren
Drug: Placebo for Aliskiren — Placebo for Aliskiren 300 mg
  Arms: Amlodipine + Placebo for Aliskiren; HCTZ + Placebo for Aliskiren; Placebo for Aliskiren + Placebo for Amlodipine; Placebo for Aliskiren + Placebo for HCTZ
Drug: Placebo for Amlodipine — Placebo for Amlodipine
  Arms: Aliskiren + Placebo for Amlodipine; Placebo for Aliskiren + Placebo for Amlodipine
Drug: Placebo for Hydrochlorothiazide (HCTZ) — Placebo for HCTZ 12.5/25 mg
  Arms: Aliskiren + Placebo for HCTZ; Placebo for Aliskiren + Placebo for HCTZ

SUMMARY:
This study was planned to provide new information regarding the role of aliskiren (with or without additional therapy with a diuretic or a Calcium channel blockers (CCB)) in elderly individuals (≥ 65 years) with systolic blood pressure (SBP) 130 to 159 mmHg, in preventing major cardiovascular (CV) events and on global measures of physical, executive and cognitive function.

DETAILED DESCRIPTION:
This was 2x2 factorial design study with 2 strata. As per protocol, the first co- Primary analysis as well as secondary analysis were aliskiren based regimen vs non-aliskiren based regimen. All aliskiren based arm were combined into the aliskiren based regimen and all non-aliskiren based arms were combined into non-aliskiren based regimen.

ELIGIBILITY:
Inclusion Criteria:

Systolic blood pressure 130 - 159 mmHg with any one of the following (1, 2 or 3):

1. Men and women aged ≥ 65 years if they have at least one of the following: (secondary prevention) Coronary heart disease

   * Previous myocardial infarction or
   * Stable angina or unstable angina with documented multi-vessel coronary artery disease, > 50% stenosis in at least 2 major coronary arteries on coronary angiography, or positive stress test (ECG or nuclear perfusion scintogram), or
   * Multi-vessel PCI, or
   * Multi-vessel CABG surgery > 4 years prior to informed consent, or with recurrent angina or ischemia following surgery Stroke/TIA Previous documented stroke or documented TIA < 1 year before informed consent Peripheral artery disease
   * Previous limb bypass surgery or percutaneous transluminal angioplasty, or
   * Previous limb or foot amputation, or
   * History of intermittent claudication, with an ankle:arm BP ratio ≤ 0.80 on at least one side, or significant peripheral artery stenosis (> 50%) documented by angiography or non-invasive testing
   * Diabetes mellitus: High-risk diabetics with evidence of end-organ damage
2. Men and women aged ≥ 65 years with no history of CVD, and with at least 1 CV risk factor (primary prevention):

   * History of dyslipidemia, defined as LDL cholesterol > 3.5 mmol/L (135 mg/dL) or HDL< 1.3 mmol/L (50 mg/dL) in women or < 1.0 mmol/L (39 mg/dL) in men or total cholesterol/HDL ratio > 5
   * History of current or recent smoking (regular tobacco use within 5 years)
   * Abdominal adiposity defined as waist/hip ratio ≥ 0.90 in women and ≥ 0.95 in men
   * History of dysglycemia defined as impaired fasting glucose (IFG - fasting plasma glucose 5.6 to 6.9 mmol/L [101 to 124 mg/dL]), or impaired glucose tolerance (IGT - fasting plasma glucose < 7 mmol/L [126 mg/dL] but 2 hour glucose 7.8 to 11.0 mmol/L [140 to 198 mg/dL]) or type 2 diabetes
   * Renal dysfunction: eGFR< 60 ml/min/1.73m2 but > 30 ml/min/1.73m2 (MDRD formula) and/or microalbuminurea/macroalbuminurea
   * Clinical evidence of left ventricular hypertrophy
3. Men and women aged ≥ 70 years if they do not have any of the above (primary prevention)

Exclusion Criteria:

1. Current treatment with aliskiren, an ACE-inhibitor, an ARB or an aldosterone antagonist and unable to discontinue this therapy in those without clinical vascular disease. Individuals with CVD or type 2 diabetes and/or renal dysfunction may receive an ACE-inhibitor or an ARB, but not both, contraindications to Aliskiren, Amlodipine or Hydrochlorothiazide.
2. Use of both thiazide diuretic and amlodipine or another calcium channel blocker. Patients on only one of these two classes of drugs are eligible
3. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg)
4. Symptomatic heart failure, requiring the use of loop diuretics
5. Hemodynamically significant primary valvular or outflow tract obstruction (e.g. aortic or mitral valve stenosis, asymmetric septal hypertrophy, malfunctioning prosthetic valve). Constrictive pericarditis. Complex congenital heart disease.
6. Acute stroke < 3 months or TIA ≤ 7 days before informed consent, acute coronary syndrome < 1 months before informed consent
7. Planned cardiac surgery or angioplasty < 3 months after informed consent or having had the procedure < 3 months before informed consent
8. Severe renal impairment eGFR ≤ 30 ml/min/1.73m2 (MDRD formula); known renal artery stenosis ; serum potassium ≥ 5.3 mmol/L
9. Chronic liver disease (i.e. cirrhosis, esophageal varices, portocaval shunt or persistent hepatitis) or abnormal liver function, i.e., alanine transaminase (ALT) or AST > 3x upper limit of normal (ULN)
10. Concurrent treatment with cyclosporine or quinidine; chronic use of non-steroidal anti-inflammatory drug (NSAIDs) or cyclooxygenase-2 (COX 2) inhibitors in patients with eGFR < 60 ml/min/1.73m2 (MDRD formula)
11. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years regardless of whether there is evidence of local recurrence or metastases
12. Other serious condition(s) likely to interfere with study participation or with the ability to complete the study. Significant psychiatric illness, senility, dementia, alcohol or substance abuse, which could impair the ability to provide informed consent and to adhere to the study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2336 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (164):
- United States (14):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Sylmar, California
  - Novartis Investigative Site, Tucker, Georgia
  - Novartis Investigative Site, Pocatello, Idaho
  - Novartis Investigative Site, Haverhill, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Westfiled, New York
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Falls Church, Virginia
  - Novartis Investigative Site, Marshfield, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (15):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Coronel Suárez, Buenos Aires
  - Novartis Investigative Site, Jenin, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Merlo, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, San Nicolás de los Arroyos, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Cipolletti, Río Negro Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, Venado Tuerto, Santa Fe Province
- Brazil (9):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Uberaba, Minas Gerais
  - Novartis Investigative Site, Campina Grande do Sul, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Marília, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Votuporanga, São Paulo
- Canada (23):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Coquitlam, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Missisauga, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Niagara Falls, Ontario
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Saint Catherines, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, St.Gorges de Beauce, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Chile (5):
  - Novartis Investigative Site, Temuco, Cautin
  - Novartis Investigative Site, Osorno, Osorno
  - Novartis Investigative Site, Vista Del Mar, Tarapacá
  - Novartis Investigative Site, Temuca, TX
  - Novartis Investigative Site, Santiago
- Colombia (16):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Manizoles, Caldas Department
  - Novartis Investigative Site, Barranquilla, Colombia
  - Novartis Investigative Site, Cali, Colombia
  - Novartis Investigative Site, Cartegena, Colombia
  - Novartis Investigative Site, Pasto, Colombia
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Cartagena, Departamento de Bolívar
  - Novartis Investigative Site, Pereira, Risaralda Department
  - Novartis Investigative Site, Floridablanca, Santander Department
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Baranquilla
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Espinal
  - Novartis Investigative Site, Montería
- Czechia (7):
  - Novartis Investigative Site, Beroun, Czech Republic
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Ústí nad Orlicí, Czech Republic
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Germany (6):
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Melsungen
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Witten
- Hungary (9):
  - Novartis Investigative Site, Komárom, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Gyöngyös
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Sopron
  - Novartis Investigative Site, Szentes
  - Novartis Investigative Site, Veszprém
- India (21):
  - Novartis Investigative Site, Adoni, Andhra Pradesh
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Bengaluru, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Wardha, Maharashtra
  - Novartis Investigative Site, Jalandhar, Punjab
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Tiruvannamalai, Tamil Nadu
  - Novartis Investigative Site, Trichy, Tamil Nadu
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Chennai
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, Nagpur
  - Novartis Investigative Site, Trichy
- Ireland (3):
  - Novartis Investigative Site, Gorey, Co. Wexford
  - Novartis Investigative Site, Ballinsloe, Galway
  - Novartis Investigative Site, Galway, Ireland
- Israel (3):
  - Novartis Investigative Site, Safed, Israel
  - Novartis Investigative Site, Giv‘atayim
  - Novartis Investigative Site, Haifa
- Malaysia (6):
  - Novartis Investigative Site, Alor Star, Kedah
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Batu Caves, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Netherlands (7):
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leiderdorp
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Velp
  - Novartis Investigative Site, Zoetermeer
- Philippines (7):
  - Novartis Investigative Site, Dasmariñas, Cavite
  - Novartis Investigative Site, Laoag, Ilocos Norte
  - Novartis Investigative Site, Quezon City, National Capital Region
  - Novartis Investigative Site, Biñan
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon City
- South Africa (4):
  - Novartis Investigative Site, Paarl, Western Province
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Pretoria
- Spain (4):
  - Novartis Investigative Site, Ferrol, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Port de Sagunt
- Sweden (5):
  - Novartis Investigative Site, Dalby
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Rättvik
  - Novartis Investigative Site, Stockholm

REFERENCES:
- [Derived] Teo KK, Pfeffer M, Mancia G, O'Donnell M, Dagenais G, Diaz R, Dans A, Liu L, Bosch J, Joseph P, Copland I, Jung H, Pogue J, Yusuf S; Aliskiren Prevention of Later Life Outcomes trial Investigators. Aliskiren alone or with other antihypertensives in the elderly with borderline and stage 1 hypertension: the APOLLO trial. Eur Heart J. 2014 Jul;35(26):1743-51. doi: 10.1093/eurheartj/ehu079. Epub 2014 Mar 9. PMID 24616335

RESULTS

PARTICIPANT FLOW:
Period: Run-in Open Label Period (4-5 Weeks)
Arm/Group | Aliskiren + Hydrochlorothiazide (HCTZ) | Aliskiren + Placebo for HCTZ | Aliskiren + Amlodipine | Aliskiren + Placebo for Amlodipine | HCTZ + Placebo for Aliskiren | Placebo for Aliskiren + Placebo for HCTZ | Amlodipine + Placebo for Aliskiren | Placebo for Aliskiren + Placebo for Amlodipine
Started | 1335 | 0 | 1001 | 0 | 0 | 0 | 0 | 0
Completed | 980 | 0 | 779 | 0 | 0 | 0 | 0 | 0
Not Completed | 355 | 0 | 222 | 0 | 0 | 0 | 0 | 0
Period: Double Blind Randomized Period
Arm/Group | Aliskiren + Hydrochlorothiazide (HCTZ) | Aliskiren + Placebo for HCTZ | Aliskiren + Amlodipine | Aliskiren + Placebo for Amlodipine | HCTZ + Placebo for Aliskiren | Placebo for Aliskiren + Placebo for HCTZ | Amlodipine + Placebo for Aliskiren | Placebo for Aliskiren + Placebo for Amlodipine
Started | 244 | 232 | 189 | 195 | 251 | 253 | 196 | 199
Completed | 242 | 229 | 188 | 191 | 247 | 245 | 190 | 196
Not Completed | 2 | 3 | 1 | 4 | 4 | 8 | 6 | 3
Not completed — Death | 1 | 1 | 1 | 2 | 1 | 5 | 2 | 1
Not completed — Withdrew informed consent/ refused visit | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 1
Not completed — Other reasons | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis Set (FAS): All randomized patients, regardless of receiving study medication.
Groups:
- Aliskiren + Hydrochlorothiazide (HCTZ): In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  Patients randomized to this arm received Aliskiren 300 mg + HCTZ 25 mg once daily.
- Aliskiren + Amlodipine: In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  Patients randomized to this arm received Aliskiren 300 mg + Amlodipine 5 mg once daily during the double blind period.
- Amlodipine + Placebo for Aliskiren: In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were run-in stratum randomized equally to the 4 arms of the Amlodipine add-on stratum.
  In double blind period, randomized patients to this arm received Amlodipine 5 mg + placebo for Aliskiren 300 mg once daily
- Total: Total of all reporting groups
Arm/Group | Aliskiren + Hydrochlorothiazide (HCTZ) | Aliskiren + Placebo for HCTZ | Aliskiren + Amlodipine | Aliskiren + Placebo for Amlodipine | HCTZ + Placebo for Aliskiren | Placebo for Aliskiren + Placebo for HCTZ | Amlodipine + Placebo for Aliskiren | Placebo for Aliskiren + Placebo for Amlodipine | Total
Number analyzed (Participants) | 244 | 232 | 189 | 195 | 251 | 253 | 196 | 199 | 1759
Age, Customized [Number; unit: participants]
  >=65 to <75 years | 165 | 174 | 127 | 125 | 180 | 189 | 135 | 134 | 1229
  >=75 years | 79 | 58 | 62 | 70 | 71 | 64 | 61 | 65 | 530
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 109 | 91 | 89 | 122 | 108 | 87 | 88 | 813
  Male | 125 | 123 | 98 | 106 | 129 | 145 | 109 | 111 | 946

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Cardiovascular Endpoints in Aliskiren Based Regimen Versus Non-Aliskiren Based Regimen
Description: The composite CV endpoint is based on the following first adjudicated events: CV death, non-fatal MI,non-fatal stroke, significant heart failure
Time Frame: End of study (209 days (median))
Population: Full Analysis set. 1759 patients were randomized as against the originally planned 11,000. A total of 25 primary CV composite endpoints had accrued during median follow-up of 209 days versus planned 2000 primary endpoints during planned follow-up of average 5 years. These low numbers significantly limit interpretation of the results.
Measure: Number; unit: participants
Groups:
- Aliskiren Based Regimen: This regimen includes all the patients who were randomized to the treatment arms that included Aliskiren such as Aliskiren + hydrochlorothiazide (HCTZ), Aliskiren + placebo for HCTZ, Aliskiren + Amlodipine, Aliskiren + placebo for Amlodipine.
- Non-Aliskiren Based Regimen: This regimen includes all the patients who were randomized to the treatment arms that did not include Aliskiren such as HCTZ + Placebo for Aliskiren, Placebo for Aliskiren + Placebo for HCTZ, Amlodipine + Placebo for Aliskiren, Placebo for Aliskiren + Placebo for Amlodipine
Arm/Group | Aliskiren Based Regimen | Non-Aliskiren Based Regimen
Number analyzed (Participants) | 860 | 899
participants | 11 | 14

2. Secondary Outcome: Change From Baseline to End of Study in Standard Assessment of Global Activities in the Elderly (SAGE) Dimensions (Part I)
Description: Decline in ability to perform everyday activities independently was measured primarily by using the Standard Assessment of Global Activities in the Elderly (SAGE) scale. The SAGE comprised of 15 questions, each describing an activity. Patient had to indicate how much difficulty he/she had encountered in performing the activity in last month. Each question's score ranges from 0 (No difficulty) to 3 (difficulty levels were mild (score = 1), moderate (score =2) and severe (score=3)). Part I of SAGE included 4 dimensions:
  * Community Cognition (maximum of scores of questions 1 to 6);
  * Instrumental Activities of daily Living (IADL) (maximum of scores of questions 7 to 10);
  * Mobility (maximum of scores of questions 11 and 12);.
  * Basic Activities of daily Living (ADL) (maximum of scores of questions 13 to 15) Each dimension's total score ranged from 0 to 3. 0=best, 3=worst A negative change in value from baseline means improvement in the ability to perform everyday activities.
Time Frame: Baseline, End of study (209 days [median])
Population: Full Analysis Set: Due to the sparse post-baseline data following early termination of the study, this analysis was not performed as planned in protocol.Hence, no meaningful conclusion could be drawn. Patients who completed both baseline and post-baseline SAGE questionnaires (Part II) were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aliskiren Based Regimen | Non-Aliskiren Based Regimen
Number analyzed (Participants) | 592 | 618
units on a scale
  Community Cognition | -0.04 (0.768) | -0.05 (0.741)
  Instrumental Activities of daily Living (IADL) | -0.06 (0.562) | -0.04 (0.505)
  Mobility | 0.01 (0.791) | 0.00 (0.779)
  ADL | -0.09 (0.525) | -0.08 (0.520)

3. Other Pre Specified Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: Mean sitting systolic blood pressure (msSBP) is the average of 2 sitting SBP measurements (2 minutes apart). Since each patient had their final follow-up visit at a different time in the trial, these measurements were classified as falling into the 6 week, 6 month, or 12 month measurement period. All available blood pressures were sorted within these periods and the last value within each time range used for analysis. At each timepoint, a patient must have both baseline and postbaseline values to be included in the analysis.
Time Frame: Baseline (BL), 6 week, 6 month and 12 month
Population: Full analysis Set : All randomized patients, regardless of receiving study medication. n=number of patients with non-missing assessments at baseline and each post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren Based Regimen | Non-Aliskiren Based Regimen
Number analyzed (Participants) | 860 | 899
mmHg
  change from Baseline to 6 week (n=821,867) | -11.9 (0.50) | -8.02 (0.48)
  change from baseline to 6 month (n=730,775) | -10.1 (0.52) | -6.8 (0.50)
  change from baseline to 12 month (n=397,399) | -7.7 (0.68) | -5.8 (0.68)

4. Primary Outcome: Number of Participants With Composite Cardiovascular Endpoints in Aliskiren+Amlodipine/HCTZ Group Versus All Placebo Group
Description: as for outcome 1
Time Frame: End of study (209 days (median))
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Aliskiren+Amlodipine/HCTZ Group: This reporting group includes all the patients who has received Aliskiren plus an additional BP lowering drug (Amlodipine or Hydrochlorothiazide). This reporting group includes patients from arms such as Aliskiren + Hydrochlorothiazide (HCTZ) and Aliskiren + Amlodipine.
- Placebo: This reporting group includes all the patients who has received placebo of aliskiren plus placebo of an additional BP lowering drug (amlodipine or hydrochlorothiazide). This reporting group includes patients from arms such as Placebo for Aliskiren + Placebo for HCTZ and Placebo for aliskiren + Placebo for Amlodipine .
Arm/Group | Aliskiren+Amlodipine/HCTZ Group | Placebo
Number analyzed (Participants) | 433 | 452
participants | 2 | 8

5. Secondary Outcome: Percentage of Participants With Standard Assessment of Global Activities in the Elderly (SAGE) Dimensions (Part II)
Description: Decline in ability to perform everyday activities independently was measured primarily by using the Standard Assessment of Global Activities in the Elderly (SAGE) scale. The SAGE was comprised of 15 questions, each describing an activity. Patient had to indicate how much difficulty he/she had encountered in performing the activity in the last month. Each question's score ranges from 0 (No difficulty) to 3 (difficulty levels were mild (score = 1), moderate (score =2) and severe (score=3)).
  Part II of SAGE included 2 dimensions:
  * "Normal" if the scores of all SAGE questions is 0 (i.e., No difficulty)
  * "Mobility Only" if scores of both SAGE questions 11 and 12 are 0
Time Frame: End of study (209 days [median])
Population: Full Analysis Set. Number of patients with all SAGE questions non-missing for the specific visit are included in this population. Due to the sparse post-baseline data following early termination of the study, this analysis was not performed as planned in protocol.Hence, no meaningful conclusion could be drawn.
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren Based Regimen | Non-Aliskiren Based Regimen
Number analyzed (Participants) | 608 | 641
percentage of participants
  Normal | 44.2 | 46.5
  Mobility Only | 66.8 | 68.6

6. Secondary Outcome: Number of Participants With Renal Dysfunction in Aliskiren Based Regimen Versus Non-Aliskiren Based Regimen
Description: The renal dysfunction (composite endpoint) was defined as the first occurrence of either of the following:
  * End-stage renal disease [ESRD] requiring dialysis or transplantation
  * Doubling of serum creatinine and reaching an eGFR < 45 ml/min/1.73 m^2.
Time Frame: End of study (209 days (median))
Population: Full Analysis set. 1759 patients were randomized as against the originally planned 11,000. The duration of study follow-up was 209 days (median) as against the planned follow-up of average 5 years. These low numbers significantly limit interpretation of the results.
Measure: Number; unit: participants
Arm/Group | Aliskiren Based Regimen | Non-Aliskiren Based Regimen
Number analyzed (Participants) | 860 | 899
participants
  ESRD requiring dialysis or transplantation | 0 | 0
  Doubling of creatinine & eGFR<45 ml/min/1.73 m^2 | 7 | 1

7. Other Pre Specified Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Mean sitting diastolic blood pressure (msDBP) is the average of 2 sitting DBP measurements (2 minutes apart). Since each patient had their final follow-up visit at a different time in the trial, these measurements were classified as falling into the 6 week, 6 month, or 12 month measurement period. All available blood pressures were sorted within these periods and the last value within each time range used for analysis. At each timepoint, a patient must have both baseline and postbaseline values to be included in the analysis.
Time Frame: Baseline (BL), 6 week, 6 month and 12 month
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren Based Regimen | Non-Aliskiren Based Regimen
Number analyzed (Participants) | 860 | 899
mmHg
  change from Baseline to 6 week (n=821,867) | -5.6 (0.31) | -3.6 (0.30)
  change from baseline to 6 month (n=730,775) | -4.9 (0.33) | -3.5 (0.32)
  change from baseline to 12 month (n=397,399) | -4.3 (0.43) | -3.9 (0.43)

8. Secondary Outcome: Number of Participants With Total Mortality in Aliskiren Based Regimen Versus Non-aliskiren Based Regimen
Description: The total mortality endpoint was defined as time to death from any cause. Total mortality analysis used the date of last follow-up including the washout period as the censoring date.
Time Frame: End of study (209 days (median))
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Aliskiren Based Regimen | Non-Aliskiren Based Regimen
Number analyzed (Participants) | 860 | 899
Participants | 5 | 9

ADVERSE EVENTS:
Description: Safety Set (SAF): The safety set consists of all randomized patients who took at least one dose of study medication. Patients were analyzed according to treatment received.
Groups:
- Run-in Period: Aliskiren + Hydrochlorothiazide (HCTZ): In run-in period (4-5 weeks) , patients on CCB background therapy and approximately 50% of patients on neither thiazide nor CCB background therapy: received Hydrochlorothiazide 12.5/25 mg and Aliskiren 150/300 mg daily in a titrated manner as per protocol.
  Patients randomized to this arm received Aliskiren 300 mg + HCTZ 25 mg once daily.
- Run-in Period: Aliskiren + Amlodipine: In run-in period (4-5 weeks) , patients on thiazide background therapy and approximately 50% of patients on neither CCB nor thiazide background therapy received Amlodipine 5 mg and Aliskiren 150/300 mg daily in a titrated manner as per protocol.
  Patients randomized to this arm received Aliskiren 300 mg + Amlodipine 5 mg once daily during the double blind period.
- Double Blind Period: Aliskiren + Hydrochlorothiazide (HCTZ): In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  Patients randomized to this arm received Aliskiren 300 mg + HCTZ 25 mg once daily.
- Double Blind Period: Aliskiren + Placebo for HCTZ: In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  In double blind period, randomized patients to this arm received Aliskiren 300 mg + placebo for HCTZ 25 mg once daily
- Double Blind Period: Aliskiren + Amlodipine: In double blind period, patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  Patients randomized to this arm received Aliskiren 300 mg + Amlodipine 5 mg once daily during the double blind period.
- Double Blind Period: Aliskiren + Placebo for Amlodipine: In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  In double blind period, randomized patients to this arm received Aliskiren 300 mg + placebo for Amlodipine 5 mg
- Double Blind Period: HCTZ + Placebo for Aliskiren: In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  In double blind period, randomized patients to this arm received HCTZ 25 mg + placebo for Aliskiren 300 mg once daily
- Double Blind Period: Placebo for Aliskiren + Placebo for HCTZ: In double blind period, all patients who successfully completed run-in with HCTZ plus Aliskiren were randomized equally to the 4 arms of the HCTZ add-on stratum.
  In double blind period, randomized patients to this arm received placebo for Aliskiren 300 mg + placebo for HCTZ 25 mg once daily
- Double Blind Period: Amlodipine + Placebo for Aliskiren: In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  In double blind period, randomized patients to this arm received Amlodipine 5 mg + placebo for Aliskiren 300 mg once daily
- Double Blind Period: Placebo for Aliskiren + Placebo for Amlod: In double blind period, all patients who successfully completed run-in with Amlodipine plus Aliskiren were randomized equally to the 4 arms of the Amlodipine add-on stratum.
  In double blind period, randomized patients to this arm received placebo for Aliskiren 300 mg + placebo for Amlodipine 5 mg once daily
Arm/Group | Run-in Period: Aliskiren + Hydrochlorothiazide (HCTZ) | Run-in Period: Aliskiren + Amlodipine | Double Blind Period: Aliskiren + Hydrochlorothiazide (HCTZ) | Double Blind Period: Aliskiren + Placebo for HCTZ | Double Blind Period: Aliskiren + Amlodipine | Double Blind Period: Aliskiren + Placebo for Amlodipine | Double Blind Period: HCTZ + Placebo for Aliskiren | Double Blind Period: Placebo for Aliskiren + Placebo for HCTZ | Double Blind Period: Amlodipine + Placebo for Aliskiren | Double Blind Period: Placebo for Aliskiren + Placebo for Amlod
Serious Adverse Events (participants affected / at risk) | 10/1335 | 10/1001 | 8/244 | 5/232 | 7/189 | 8/195 | 4/251 | 6/253 | 3/196 | 7/199
Other Adverse Events (participants affected / at risk) | 7/1335 | 19/1001 | 6/244 | 5/232 | 9/189 | 8/195 | 6/251 | 5/253 | 14/196 | 3/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: Aliskiren + Hydrochlorothiazide (HCTZ) (N=1335) | Run-in Period: Aliskiren + Amlodipine (N=1001) | Double Blind Period: Aliskiren + Hydrochlorothiazide (HCTZ) (N=244) | Double Blind Period: Aliskiren + Placebo for HCTZ (N=232) | Double Blind Period: Aliskiren + Amlodipine (N=189) | Double Blind Period: Aliskiren + Placebo for Amlodipine (N=195) | Double Blind Period: HCTZ + Placebo for Aliskiren (N=251) | Double Blind Period: Placebo for Aliskiren + Placebo for HCTZ (N=253) | Double Blind Period: Amlodipine + Placebo for Aliskiren (N=196) | Double Blind Period: Placebo for Aliskiren + Placebo for Amlod (N=199)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug interaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral hypoperfusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: Aliskiren + Hydrochlorothiazide (HCTZ) (N=1335) | Run-in Period: Aliskiren + Amlodipine (N=1001) | Double Blind Period: Aliskiren + Hydrochlorothiazide (HCTZ) (N=244) | Double Blind Period: Aliskiren + Placebo for HCTZ (N=232) | Double Blind Period: Aliskiren + Amlodipine (N=189) | Double Blind Period: Aliskiren + Placebo for Amlodipine (N=195) | Double Blind Period: HCTZ + Placebo for Aliskiren (N=251) | Double Blind Period: Placebo for Aliskiren + Placebo for HCTZ (N=253) | Double Blind Period: Amlodipine + Placebo for Aliskiren (N=196) | Double Blind Period: Placebo for Aliskiren + Placebo for Amlod (N=199)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 7 | 0 | 1 | 4 | 0 | 0 | 2 | 7 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 7 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 5 | 4 | 3 | 6 | 2 | 4 | 1 | 5 | 1

LIMITATIONS AND CAVEATS:
Due to early termination, 1759 patients were randomized as against 11,000. Only 25 primary endpoints had accrued during median follow-up of 209 days as against planned 2000 in 5 years. These low numbers significantly limit interpretation of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.